CLINICAL TRIAL: NCT00400101
Title: A Randomized Placebo-Controlled Phase Ia Malaria Vaccine Trial of Two Virosome-Formulated Synthetic Peptides in Healthy Adult Volunteers
Brief Title: Phase Ia Malaria Vaccine Trial of Two Virosome-Formulated Peptides
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEV001
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Falciparum Malaria
Keywords: Malaria; Vaccine; Plasmodium; falciparum; Phase I; Peptide; Virosome; safety; immunogenicity
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Malaria Vaccines

INTERVENTIONS:
Biological: Virosome-formulated synthetic peptides (malaria vaccine)

SUMMARY:
Influenza virosomes represent an innovative human-compatible antigen delivery system that has already proven its suitability for subunit vaccine design. The aim of the study was to proof the concept that virosomes can also be used to elicit high titers of antibodies against synthetic peptides derived from the circumsporozoite protein and from the apical-membrane-antigen 1 and that the formulations are safe in humans.

DETAILED DESCRIPTION:
Influenza virosomes represent an innovative human-compatible antigen delivery system that has already proven its suitability for subunit vaccine design. The aim of the study was to proof the concept that virosomes can also be used to elicit high titers of antibodies against synthetic peptides. The specific objective was to demonstrate the safety and immunogenicity of two virosome-formulated P. falciparum protein derived synthetic peptide antigens given in two different doses alone or in combination.

Methodology The design was a single blind, randomized, placebo controlled, dose-escalating study involving 46 healthy Caucasian volunteers aged 18-45 years. Five groups of 8 subjects received virosomal formulations containing 10 ug or 50 ug of AMA 49-CPE, an apical membrane antigen-1 (AMA-1) derived synthetic phospatidylethanolamine (PE)-peptide conjugate or 10 ug or 50 ug of UK39, a circumsporozoite protein (CSP) derived synthetic PE-peptide conjugate or 50 ug of both antigens each. A control group of 6 subjects received unmodified virosomes. Virosomal formulations of the antigens (designated PEV301 and PEV302 for the AMA-1 and the CSP virosomal vaccine, respectively) or unmodified virosomes were injected i. m. on days 0, 60 and 180.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes, aged between 18 and 45 years, with a BMI > 18.5 and <30 were included if they gave written informed consent

Exclusion Criteria:

* Chronix or acute illness, immunosuppression, lived in the past in a malaria endemic area, had visited such an area in the last 12 months, or had a history of clinical malaria

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2003-11; Study Completion 2005-10

PRIMARY OUTCOMES:
Incidence of adverse events
Antibody concentration by Elisa

SECONDARY OUTCOMES:
Antibody concentration by IFAT and Western blot
Cellular immunity

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD PhD, Principal Investigator — Swiss Tropical & Public Health Institute

REFERENCES:
- [Derived] Okitsu SL, Silvie O, Westerfeld N, Curcic M, Kammer AR, Mueller MS, Sauerwein RW, Robinson JA, Genton B, Mazier D, Zurbriggen R, Pluschke G. A virosomal malaria peptide vaccine elicits a long-lasting sporozoite-inhibitory antibody response in a phase 1a clinical trial. PLoS One. 2007 Dec 5;2(12):e1278. doi: 10.1371/journal.pone.0001278. PMID 18060072
- [Derived] Genton B, Pluschke G, Degen L, Kammer AR, Westerfeld N, Okitsu SL, Schroller S, Vounatsou P, Mueller MM, Tanner M, Zurbriggen R. A randomized placebo-controlled phase Ia malaria vaccine trial of two virosome-formulated synthetic peptides in healthy adult volunteers. PLoS One. 2007 Oct 10;2(10):e1018. doi: 10.1371/journal.pone.0001018. PMID 17925866